CLINICAL TRIAL: NCT06419582
Title: A Phase 2/3, Multicenter, Inpatient, Placebo-Controlled, Double-blind Trial of BHV-7000 for the Acute Treatment of Manic Episodes, With or Without Mixed Features, Associated With Bipolar I Disorder
Brief Title: BHV-7000 Acute Treatment of Bipolar Mania
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biohaven Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Organization: Biohaven Pharmaceuticals, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BHV7000-204
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: bipolar; mania; manic episode; manic state; bipolar disorder type 1; manic depressive; manic bipolar; mixed features; mixed episode; mixed mania; bipolar episode
MeSH Terms: conditions — Bipolar Disorder; Mania

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BHV-7000 (Experimental)
  Interventions: Drug: BHV-7000
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BHV-7000 — BHV-7000 75 mg taken once daily for 21 days
  Arms: BHV-7000
Drug: Placebo — Matching placebo taken once daily for 21 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether BHV-7000 is a safe and effective acute treatment for manic episodes in bipolar disorder I.

ELIGIBILITY:
Key Inclusion Criteria:

1. Participant must be voluntarily hospitalized for a current manic episode.
2. Male and female participants 18 years to 75 years of age at the time of the screening visit.
3. Body Mass Index (BMI) must be ≥ 18 kg/m2 and ≤ 35 kg/m2.
4. Meets DSM-5 criteria for bipolar disorder type I, with or without mixed features, as confirmed by MINI interview with at least one well- defined prior mood episode (in addition to the current episode). The most recent prior manic episode must have occurred in the last 2 years.
5. Episode of mania must not exceed 12 weeks in duration.
6. Participants must be able and willing to discontinue all other psychotropic medications during the Screening Phase (e.g., antidepressant, antimanic, antipsychotic medications).

Key Exclusion Criteria:

1. Rapid cycling is excluded as defined herein by subjects who have experienced ≥ 6 distinct mood episodes in a year. Consecutive mood episodes must be demarcated either by a partial or full remission of at least 2 months' duration or by a switch to an episode of opposite polarity. Each manic or mixed episode must have lasted at least 1 week, and each hypomanic episode must have lasted at least 4 days.
2. Participants with a confirmed lifetime history of schizophrenia, psychotic disorders, dementia, delirium, amnesia, neurodegenerative disease, traumatic brain injury with clinically significant sequalae, seizure disorder, or other neurocognitive disorder. Previous diagnosis of psychotic spectrum disorders are allowable if the Investigator deems the diagnosis to be describing symptoms related to bipolar disorder.
3. Any medical condition, based on the judgement of the Investigator, that would confound the ability to adequately assess safety and efficacy outcome measures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2024-05-28 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Young Mania Rating Scale (YMRS) total score from baseline to day 21 | Baseline (day 1) to day 21
  The YMRS is a clinician administered scale that consists of 11 items used to assess the subject's symptoms of mania (total scores range from 0 to 60). The higher the YMRS score, the more severe the subject's symptoms of mania.

SECONDARY OUTCOMES:
Change in Clinical Global Clinical Impression - Severity Scale (CGI-S) total score | Baseline (day 1) to day 21
  This objective will be measured by the change in Clinical Global Impression of Severity (CGI-S) score from baseline (day 1) to day 21). The CGI-S is a global index of patient disease severity as rated by the clinician on a scale from 1 to 7, where 7 represents most severe patients.
Percentage of participants showing treatment response | Baseline (day 1) to day 21
  Treatment response is defined as greater than or equal to 50% reduction from baseline to day 21 on the YMRS total score.
  The YMRS is a clinician administered scale that consists of 11 items used to assess the subject's symptoms of mania (total scores range from 0 to 60). The higher the YMRS score, the more severe the subject's symptoms of mania.
Percentage of participants showing treatment remission | Baseline (day 1) to day 21
  Treatment remission is defined as score of less than or equal to 12 on the YMRS total score from baseline to day 21.
  The YMRS is a clinician administered scale that consists of 11 items used to assess the subject's symptoms of mania (total scores range from 0 to 60). The higher the YMRS score, the more severe the subject's symptoms of mania.
Change in Young Mania Rating Scale (YMRS) total score from baseline to day 7 | Baseline (day 1) to day 7
  This objective will be measured by the change in YMRS total score from baseline (day 1) to day 7. The YMRS is a clinician administered scale that consists of 11 items used to assess the subject's symptoms of mania (total scores range from 0 to 60).
  The higher the YMRS score, the more severe the subject's symptoms of mania.
Change in Young Mania Rating Scale (YMRS) total score from baseline to day 4 | Baseline (day 1) to day 4
  This objective will be measured by the change in YMRS total score from baseline (day 1) to day 4. The YMRS is a clinician administered scale that consists of 11 items used to assess the subject's symptoms of mania (total scores range from 0 to 60).
  The higher the YMRS score, the more severe the subject's symptoms of mania.
Change in Montgomery-Åsberg Depression Rating Scale (MADRS) score from baseline to day 21 | Baseline (day 1) to day 21
  This objective will be measured by the change in MADRS total score from baseline (day 1) to day 21. The MADRS, Montgomery-Asberg Rating Scale, measures depression on a 10 item scale. The overall score ranges from 0 to 60. The higher the MADRS score indicates more severe depression.
Number of Participants With Serious AEs (SAEs), AEs Leading to Study Drug Discontinuation, and AEs judged to be related to study medication | Baseline (day 1) to day 21
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with SAEs, AEs leading to discontinuation, AEs judged to be related to study medication that are observed during the Double-blind Treatment Phase (21 days).
Number of Participants With Clinically Significant Laboratory Abnormalities | Baseline (day 1) to day 21
  To assess the safety and tolerability of BHV-7000. This objective will be measured by assessing the number of unique subjects with grade 3 or 4 laboratory abnormalities.
Number of Participants With Vital Sign Abnormalities | Baseline (day 1) to day 21
Number of Participants With Electrocardiogram (ECG) Abnormalities specific to QTc elevation | Baseline (day 1) to day 21

CONTACTS AND LOCATIONS:
Locations (32):
- United States (32):
  - Pillar Clinical Research, LLC, Bentonville, Arkansas
  - WIRG, Little Rock, Arkansas
  - WRN, Rogers, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - CIT LA, Bellflower, California
  - ProScience Research Group, Culver City, California
  - Cenexel CNS, Garden Grove, California
  - Synergy San Diego, Lemon Grove, California
  - NRC Research Institute, Orange, California
  - CIT IE, Riverside, California
  - Cenexel CNS, Torrance, California
  - Segal Trials - Larkin Behavioral Health Services-Inpatient & Early Phase Site, Hollywood, Florida
  - Cenexel - RCA, Hollywood, Florida
  - LCC Medical Research Inst, Miami, Florida
  - Floridian Neuroscience Institute, Miami Lakes, Florida
  - Segal Trials - Miami Lakes Medical Research-Inpatient & Early Phase Site, Miami Lakes, Florida
  - Neuroscience Research Institute, West Palm Beach, Florida
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - CenExel iResearch, LLC, Decatur, Georgia
  - CenExel iResearch, LLC, Savannah, Georgia
  - Uptown Research Institute, Chicago, Illinois
  - Pillar Clinical Research, Chicago, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Precise Clinical Research, Flowood, Mississippi
  - Arch Clinical Trials, St Louis, Missouri
  - Hassman Research Institute, Marlton, New Jersey
  - RBA, Staten Island, New York
  - Midwest Clinical Research Center, Dayton, Ohio
  - NBCR, North Canton, Ohio
  - Community Clinical Research, Inc., Austin, Texas
  - InSite Clinical Research, LLC, DeSoto, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas